CLINICAL TRIAL: NCT03823820
Title: Bioimpedance In Pregnancy and Labour: A Fluid Balance Concept Study.
Acronym: BiPAL
Status: Recruiting | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: Edge ID 120909
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hydration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cesarean section: Women attending for elective CS.
  Interventions: Other: Bioimpedance Analyser
- Induction of labour: Women admitted for induction of labour and expected to stayed in hospital for more than 24 hours.
  Interventions: Other: Bioimpedance Analyser
- pregnancy complication group: Maternal condition that could affect body fluid including:
  * Pre-eclampsia requiring hospital admission.
  * Hyperemesis gravidarum.
  * Major postpartum haemorrhage.
  Interventions: Other: Bioimpedance Analyser
- control: Gestational age matched controls.
  Interventions: Other: Bioimpedance Analyser

INTERVENTIONS:
Other: Bioimpedance Analyser — Bio-electrical impedance analysis (BIA) measures whole body (or regional) impedance by means of an electric current transmitted at different frequencies.

SUMMARY:
The purpose of our study is to find out if using a simple bed side test can tell us information about changes that occur in women's body water content. We would like to check if certain medical conditions could affect body water contents.

DETAILED DESCRIPTION:
Maternal cardiovascular physiology evolves during the course of pregnancy to accommodate the growing foetus. In order that the uterine artery can deliver 10% of the entire maternal cardiac output, there are considerable structural and physiological changes that take place. There is a 30% increase in global arterial compliance, predominantly due to vasodilation at the level of the renal arteries, which leads to a reduced total peripheral resistance. Stroke volume increases due to the plasma expansion and increasing total blood volume. All water compartments show an absolute and relative increase with advancing gestation and eventually water represents the largest component of weight gain in pregnancy. These changes have been measured and known to clinicians for decades. Yet, it is only in the recent past, that the possible clinical relevance of assessing total body water and extracellular body water has been enhanced by the cross over of hypertensive disorders of pregnancy with obesity epidemics.

Bio-electrical impedance analysis (BIA) measures whole body (or regional) impedance by means of an electric current transmitted at different frequencies. New techniques allow measurement of total body water with separation into extracellular and intracellular water. Current evidence suggests that BIA may provide useful information not only in different well-established patient groups (renal dialysis, malnutrition), but also in critically ill patients with burns, trauma and sepsis undergoing fluid resuscitation.

There are a limited number of studies assessing the use of BIA during pregnancy. In a longitudinal study of 126 pregnant women, Piuri and colleagues assessed changes of bio-impedance analysis among low-risk pregnant woman recruited in the first trimester and followed their progress. They found that women who developed hypertensive disorders of pregnancy (HDP) showed significantly different bioimpedance from control cases. Total Body Water (TBW)indices were highly significantly different from the first trimester. In pregnancies delivered of small for gestational age (SGA) newborns, these indices were the opposite of the values observed in patients with HDP-average for gestational age (AGA).TBW in these patients was significantly reduced compared with normal pregnancies. The authors concluded that the bioelectrical impedance is a fast, simple, noninvasive way to assess the TBW content in pregnancy and bio-impedance might help to identify, early in gestation, patients at risk of developing different clinical phenotypes of hypertensive disease of pregnancy and SGA fetuses.

In a prospective observational study of 3000 pregnant women, Kent and colleagues examined the use of multi frequency segmental bioelectric impedance analysis in the first trimester of pregnancy for assessment of maternal body composition as predictors of increased birth weight. They observed that on direct measurements of body composition, birth weight correlated positively with maternal fat-free mass and not adiposity.

Several factors may influence the progression of normal labour. It has been postulated that the routine administration of intravenous fluids to keep women adequately hydrated during labour may reduce the period of contraction and relaxation of the uterine muscle, and may ultimately reduce the duration of the labour. It has also been suggested that intravenous fluids may reduce caesarean section rates (CS) for prolonged labour. Conversely, excessive volumes of intravenous fluids may pose risks to both the mother and her new-born with different fluids being associated with different risks.

In a Cochrane systematic review, Dawood and colleagues reported that administration of intravenous fluids compared with oral intake alone demonstrated a reduction in the duration of labour. The findings of other trials suggested that if a policy of no oral intake is applied, then the duration of labour in nulliparous women may be shortened by the administration of intravenous fluids at a rate of 250 ml/hour rather than 125ml/hour. However, there was no objective assessment of hydration status.

However, the benefits of routine administration of intravenous fluids to labouring women has not been adequately elucidated although it is a widely-adopted policy, and there is no consensus on the type or volume of fluid that are required, or indeed, whether intravenous fluids are at all necessary. Women may be able to adequately hydrate themselves if they were allowed oral fluids during labour.

Enhanced recovery was initially introduced for patients having minimally-invasive laparoscopic surgery. Following its introduction in colorectal surgery, it is now advocated for many other specialities including Obstetrics. Enhanced recovery has transformed the delivery of perioperative practice. The core ethos of enhanced recovery is to speed up a patient's recovery after surgery and improve patient outcomes, with associated benefits for staff and healthcare systems.

Patients are given clear instructions about fluid and food intake before the operation. Currently there is limited data about hydration state at the time of admission for operation. Women having their operation on the morning of admission are advised to follow the following instructions: a) they should not eat food after 0200h. b) They can drink water until 0600h. c) At 0600h women should consume 400ml (2x 200ml bottles supplied at outpatient 'pre-clerking' clinic) of high energy carbohydrate drink before they attend hospital. Women should then remain nil by mouth, unless advised differently by the hospital team. Ranitidine and all routine medications (unless directed otherwise on the intrapartum care plan) should be taken at 0600h. Women having operations in the afternoon are advised a) to have light breakfast such as cereal, toast and fruit. b) Women should not eat food after 0600h but may drink water until 1000h.

Hypertensive disorders during pregnancy carry risks for the mother and the baby and it is one of the leading causes of maternal morbidity and mortality death in the worldwide. A UK study reported that one-third of severe maternal morbidity was a consequence of hypertensive conditions and a study conducted in the USA found that over half of admissions for acute kidney failure, one-quarter of admissions for coagulopathy and nearly one-third of admissions for ventilation or cerebrovascular disorders occurred in women with hypertensive disorders.

In a semi-longitudinal cohort study from Italy, Wilfried and colleagues examined changes in body fluid composition using Bioimpedance analyser of women with early onset preeclampsia (75 subjects) and late onset preeclampsia (117 subjects) and compared results to healthy controls. They observed significant difference in extracellular water among women with preeclampsia across trimesters. However, changes in body fluid and degree of severity of pre-eclampsia were not examined before. Other conditions that could affect body composition of water during pregnancy includes hyperemesis gravidarum, poor renal or cardiac function, major postpartum haemorrhage, and sepsis.

ELIGIBILITY:
Inclusion Criteria: pregnant women at age of 16 or over with a viable pregnancy and who will fulfil the following:

* Group I: Women attending for elective CS.
* Group II: Women admitted for induction of labour and expected to stay stay in hospital for more than 24 hours.
* Group III: Maternal condition that could have direct impact on body fluid including:

  1. Pre-eclampsia requiring hospital admission.
  2. Hyperemesis gravidarum requiring hospital admission.
  3. Major postpartum haemorrhage (equal or greater than 1000 ml following delivery).
* Group IV: gestational age matched controls.

Exclusion criteria:

* Maternal age less than 16 years at booking.
* Women who are not capable of giving consent.
* Women with learning disabilities/difficulties.
* Unable to speak or read English to the appropriate level.
* Prisoners.
* Any others deemed to belong to a vulnerable group.
* Women who require pace maker or defibrillators.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women admitted for caesarean section, induction of labour or has a medical condition that affect amount of fluid inside the body.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2029-02-14 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Bioimpedance assessment of hydration status | on admission
  assessment of extracellular and intra-cellular body fluid using Bio-electrical impedance analysis and comparing results to standard fluid chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Univercity Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Background] McCARTNEY CP, POTTINGER RE, HARROD JP Jr. Alterations in body composition during pregnancy. Am J Obstet Gynecol. 1959 May;77(5):1038-53. doi: 10.1016/0002-9378(59)90048-1. No abstract available. PMID 13649774
- [Background] HUTCHINSON DL, PLENTL AA, TAYLOR HC Jr. The total body water and the water turnover in pregnancy studied with deuterium oxide as isotopic tracer. J Clin Invest. 1954 Feb;33(2):235-41. doi: 10.1172/JCI102890. No abstract available. PMID 13130691
- [Background] Pirani BB, Campbell DM, MacGillivray I. Plasma volume in normal first pregnancy. J Obstet Gynaecol Br Commonw. 1973 Oct;80(10):884-7. doi: 10.1111/j.1471-0528.1973.tb02146.x. No abstract available. PMID 4585824
- [Background] Piuri G, Ferrazzi E, Bulfoni C, Mastricci L, Di Martino D, Speciani AF. Longitudinal changes and correlations of bioimpedance and anthropometric measurements in pregnancy: Simple possible bed-side tools to assess pregnancy evolution. J Matern Fetal Neonatal Med. 2017 Dec;30(23):2824-2830. doi: 10.1080/14767058.2016.1265929. Epub 2016 Dec 14. PMID 27892802
- [Background] Kent E, O'Dwyer V, Fattah C, Farah N, O'Connor C, Turner MJ. Correlation between birth weight and maternal body composition. Obstet Gynecol. 2013 Jan;121(1):46-50. doi: 10.1097/aog.0b013e31827a0052. PMID 23232753
- [Background] Dawood F, Dowswell T, Quenby S. Intravenous fluids for reducing the duration of labour in low risk nulliparous women. Cochrane Database Syst Rev. 2013 Jun 18;2013(6):CD007715. doi: 10.1002/14651858.CD007715.pub2. PMID 23780639
- [Background] The Association of Anaesthetists of Great Britain and Ireland Obstetric Anaesthetists' Association (2000). OAA/AAGBI Guidelines for Obstetric Anaesthetic Services Revised Edition 2005. London: The Association of Anaesthetists of Great Britain and Ireland Obstetric Anaesthetists' Association.
- [Background] The Association of Anaesthetists of Great Britain and Ireland. Immediate Postanaesthetic Recovery. September 2002. www.aagbi.org.
- [Background] NICE Advice QP Case Study Published November 2009 Last updated May 2016
- [Background] DOH Nov 2009. Enhanced Recovery for Elective Surgery. www.evidence.nhs.uk/qualityand productivity
- [Background] Gregory, R et al. Can pre-operative carbohydrate loading be used in diabetic patients undergoing colorectal surgery? British Journal of Diabetes. 2011: Vol 14-3. P102-4.
- [Background] Management of adults with diabetes undergoing surgery and elective procedures: Improving standards (revised 2016). The Joint British Diabetes Societies for inpatient care. Diabetes UK.
- [Background] Enhanced Recovery for Elective Caesarean Sections. University of Leicester Working Party. Guideline Register No: C15/2017.
- [Background] Knight M; UKOSS. Eclampsia in the United Kingdom 2005. BJOG. 2007 Sep;114(9):1072-8. doi: 10.1111/j.1471-0528.2007.01423.x. Epub 2007 Jul 6. PMID 17617191
- [Background] Lyons G. Saving mothers' lives: confidential enquiry into maternal and child health 2003-5. Int J Obstet Anesth. 2008 Apr;17(2):103-5. doi: 10.1016/j.ijoa.2008.01.006. Epub 2008 Mar 4. No abstract available. PMID 18308550
- [Background] Schutte JM, Schuitemaker NW, van Roosmalen J, Steegers EA; Dutch Maternal Mortality Committee. Substandard care in maternal mortality due to hypertensive disease in pregnancy in the Netherlands. BJOG. 2008 May;115(6):732-6. doi: 10.1111/j.1471-0528.2008.01702.x. PMID 18410657
- [Background] Waterstone M, Bewley S, Wolfe C. Incidence and predictors of severe obstetric morbidity: case-control study. BMJ. 2001 May 5;322(7294):1089-93; discussion 1093-4. doi: 10.1136/bmj.322.7294.1089. PMID 11337436
- [Background] Kuklina EV, Ayala C, Callaghan WM. Hypertensive disorders and severe obstetric morbidity in the United States. Obstet Gynecol. 2009 Jun;113(6):1299-1306. doi: 10.1097/AOG.0b013e3181a45b25. PMID 19461426
- [Background] Gyselaers W, Vonck S, Staelens AS, Lanssens D, Tomsin K, Oben J, Dreesen P, Bruckers L. Body fluid volume homeostasis is abnormal in pregnancies complicated with hypertension and/or poor fetal growth. PLoS One. 2018 Nov 1;13(11):e0206257. doi: 10.1371/journal.pone.0206257. eCollection 2018. PMID 30383796